CLINICAL TRIAL: NCT01118416
Title: Risk Reduction Intervention for Vulnerable Young Adult Males
Acronym: YMHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Jeffrey T. Parsons, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA020366 (NIH)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Sex; Substance Use; HIV
Keywords: sexual risk; substance use; HIV; prevention; intervention; Motivational Enhancement Therapy; young men who have sex with men
MeSH Terms: conditions — Coitus; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention condition (Experimental): Participants randomized to the intervention condition will undergo 4 one-hour sessions of motivational interviewing (MI), during which their sexual risk taking and substance use patterns will be discussed with a trained counselor with the goal of reducing instances of unprotected anal sex and substance use.
  Interventions: Behavioral: HIV prevention intervention randomized control trial
- Education condition (Active Comparator): Participants randomized to the education condition will undergo 4 one-hour sessions during which they will view video segments and discuss sexual risk taking and substance use with a health educator, with the goal of reducing instances of unprotected anal sex and substance use by making informed decisions.
  Interventions: Behavioral: HIV prevention intervention randomized control trial

INTERVENTIONS:
Behavioral: HIV prevention intervention randomized control trial — Substance using HIV-negative young MSM who engage in sexual risk are randomized to either a motivational interviewing or an education condition to reduce sexual risk and drug use.

SUMMARY:
The primary aim of this study is to test a brief 4-session risk reduction intervention, based on Motivational Enhancement Therapy (MET) to reduce the co-occurrence of club drug use and sexual risk taking behaviors among non-treatment seeking young men who have sex with men (YMSM) in NYC.

DETAILED DESCRIPTION:
This study is a randomized clinical trial. A sample of 300 non-treatment seeking YMSM (ages 18-24) who report risky sex and club drug use in the past 90 days are being enrolled using active and passive community-based recruitment strategies in NYC. After baseline assessment, participants are being randomly assigned to one of two study arms: a Brief Risk Reduction Intervention Condition - a four session MET intervention piloted for feasibility and acceptability among YMSM, designed to increase readiness to change club drug use and unprotected sex; or an Education Comparison Condition - four sessions of facilitated education regarding the effects of club drugs and unprotected sex. Participants undergo follow-up assessments 3, 6, 9, and 12 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 days of drug use (cocaine, ketamine, ecstasy, methamphetamine, or GHB) in the past 90 days;
* At least 1 instance of unprotected anal sex in the past 90 days;
* Biological male;
* HIV-negative;
* Residential stability;
* Ability to communicate in written English.

Exclusion Criteria:

* Unstable, serious psychiatric symptoms;
* Currently suicidal/homicidal;
* Evidence of gross cognitive impairment;
* Reports current enrollment in a drug or HIV related intervention or research study.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2006-06; Primary Completion 2010-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Sexual risk | every three months over the course of a year
  Participants in the MET condition will report greater reductions in the number of unprotected anal intercourse acts and in the proportion of days of club drug use than those in the education comparison condition at the end of the intervention period (3 months) and will maintain greater reductions in the number of unprotected anal intercourse acts and the proportion of days of club drug use than those in the education comparison condition at the three follow-up assessments (6, 9, and 12 months).

SECONDARY OUTCOMES:
motivation to change club drug use and unsafe sex over 12 months | every three months over the course of a year
  The following factors assessed at baseline will predict club drug use and unsafe sex over the 12-month outcome period: baseline severity of club drug use, baseline severity of other substance use, motivation, decisional balance, and self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Parsons, PhD, Principal Investigator — Hunter College of CUNY and Center for HIV/AIDS Educational Studies and Training
Locations (1):
- Center for HIV/AIDS Educational Studies and Training of Hunter College, CUNY, New York, New York, United States

REFERENCES:
- See also: Center for HIV/AIDS Educational Studies and Training website — http://www.hunter.cuny.edu/chest/